CLINICAL TRIAL: NCT03171415
Title: A Double Blind, Randomized, Placebo Controlled, Dose Escalation Phase 2a Clinical Trial for the Evaluation of Safety, Efficacy and Thermogenesis-induction of RZL-012 in Overweight and Obese Volunteers
Brief Title: Evaluation of Safety, Efficacy and Thermogenesis-induction of RZL-012 in Overweight and Obese Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RZL-012-P2aUS-001
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Weight Loss; Overweight and Obesity
Keywords: Obesity; Overweight; Thermogenesis; Fat reduction
MeSH Terms: conditions — Obesity; Weight Loss; Overweight | interventions — RZL-012

STUDY DESIGN:
Intervention Model Description: This is a consecutive 4 cohort, dose escalation placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind, Randomized, Placebo Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RZL-012 (Experimental): A single-time injection, multiple subcutaneous injections of RZL-012 administered into 8-36 sites (0.1mL per site):
  1. 40mg RZL-012 -administered at 8 sites
  2. 80mg RZL-012 - administered at 16 sites
  3. 120mg RZL-012 - administered at 24 sites
  4. 180mg RZL-012 - administered at 36 sited
  Interventions: Drug: RZL-012
- Placebo (Placebo Comparator): A single-time injection, multiple subcutaneous injections of Placebo administered into 8-36 sites (0.1mL per site)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RZL-012 — Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 8-36 sites (0.1mL per site) into the abdominal subcutaneous fat.
  Arms: RZL-012
Drug: Placebo — Subject receive a single-time injection. Multiple injections of the Placebo are administered at 8-36 sites (0.1mL per site) into the abdominal subcutaneous fat.
  Arms: Placebo

SUMMARY:
Obesity is a direct result of food-intake in excess of body energy expenditure. Thus, induction of increased energy expenditure via the activation of thermogenesis at targeted anatomical sites can counterbalance obesity. This trial aims to study RZL-012, a novel compound, in treating obesity by activating thermogenesis in subcutaneous fat.

DETAILED DESCRIPTION:
Obesity is a direct result of food-intake in excess of body energy expenditure. Therefore, a feasible approach to combat obesity is via energy-consuming activities, such as physical exercise. Unfortunately, our modern society is moving in the other direction, spending more time in immobilized positions, at work and at home. An alternative strategy for the induction of increased energy expenditure is via the activation of thermogenic cells that utilize fat to produce heat.RZL-012 is a novel molecule that enables de-novo generation of thermogenic tissue at favorable anatomical sites. As a result, the extra fat accumulated in obese persons will be turned into heat. This is a double blind, randomized, placebo controlled, dose escalation Phase 2a clinical trial for the evaluation of safety, efficacy and thermogenesis-induction of RZL-012 in overweight and obese volunteers. This trial aims to study the ability of RZL-012 in treating obesity via the induction of thermogenic foci in subcutaneous fat.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male subjects, 20-60 years old.
2. Subject is considered overweight and obese, with 27.5 < BMI ≤ 34.9.
3. Significant subcutaneous abdominal fat as defined by Waist to hip ratio (WHR) ≥ 0.9.
4. Subjects with stable weight in the last 3 months by medical history.
5. Not one of the following eating disorders by subject's declaration: anorexia nervosa, bulimia nervosa.
6. Generally considered healthy according to medical history, physical examination, electrocardiogram (ECG) and laboratory evaluation with a special emphasis on metabolic parameters (fasting glucose concentration < 100 mg, normal blood pressure).
7. Subject is willing to refrain from sexual activity or agrees to use a double-barrier contraceptive device (e.g., condom and spermicide) for 4 weeks after treatment with RZL 012.
8. Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
9. Subjects must sign an informed consent indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

1. Subjects weighing less than 75 kg.
2. Subjects who have reduced/gained weight more than 5% of their current body weight in the last 3 months.
3. Unable to tolerate subcutaneous injection.
4. Subjects with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorders, that in the opinion of the investigator put the subject at significant risk, are not eligible.
5. Subjects who test positive to either Hepatitis B virus (HBV), Hepatitis C virus (HCV), or Human immunodeficiency virus (HIV) are not eligible.
6. Subjects with a clinical history of primary or secondary immunodeficiency, autoimmune disease or subjects taking immunosuppressive drugs such as corticosteroids are ineligible.
7. As a result of medical review, physical examination, the PI (or medically qualified nominee) considers the subject unfit for the study.
8. Medication use on regular basis.
9. Positive drug and alcohol tests.
10. Known sensitivity to components of the injection formulation.
11. Prior wound, tattoo or infection in the treated area.
12. Excessive growth of hair in the abdomen region.
13. Claustrophobia or MRI incompatible device or implant.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was designed to enroll 32 subjects. In practice, 33 subjects were enrolled into the study. In cohort 3, one subject that was injected with plcebo was lost to follow up 3 days following injection. Therefore, an additional subject was enrolled and injected with placebo but he also was lost to follow up, 7 days following injection.
Groups:
- RZL-012 Cohort 1: A single-time injection, multiple subcutaneous injections of 40mg RZL-012 administered into 8 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 8 (0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 2: A single-time injection, multiple subcutaneous injections of 80 mg RZL-012 administered into 16 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 16 (0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 3: A single-time injection, multiple subcutaneous injections of 120 mg RZL-012 administered into 24 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 24 (0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 4: A single-time injection, multiple subcutaneous injections of 180 mg RZL-012 administered into 36 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 36 (0.1mL per site) into the abdominal subcutaneous fat.
- Placebo: A single-time injection, multiple subcutaneous injections of Placebo administered into 8/16/24/36 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of Placebo are administered at 8/16/24/36 (0.1mL per site) into the abdominal subcutaneous fat.
Period: Overall Study
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Started | 6 | 6 | 6 | 6 | 9
Completed | 6 | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 20-60 years old, overweight and obese by BMI definition (27.5 < BMI ≤ 34.9), adult males.
Groups:
- RZL-012 Cohort 2: A single-time injection, multiple subcutaneous injections of 80mg RZL-012 administered into 16 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 16(0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 3: A single-time injection, multiple subcutaneous injections of 120mg RZL-012 administered into 24 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 24(0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 4: A single-time injection, multiple subcutaneous injections of 180mg RZL-012 administered into 36 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 36(0.1mL per site) into the abdominal subcutaneous fat.
- Placebo: A single-time injection, multiple subcutaneous injections of Placebo administered into 8/16/24/36 sites (0.1mL per site)
  Placebo: Subject receive a single-time injection. Multiple injections of the Placebo are administered at8/16/24/36 (0.1mL per site) into the abdominal subcutaneous fat.
- Total: Total of all reporting groups
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 9 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (2.1) | 44.5 (12.1) | 40 (11.8) | 41.7 (13.2) | 39.2 (10.3) | 39.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 9 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 5 | 6 | 6 | 8 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Safety: The Incidence of Treatment-related Adverse Events [AEs]
Description: AEs will be assessed by significant clinical changes in safety parameter (e.g. vital signs, ECG, clinical laboratory evaluations)AEs incidence will be by body system, seriousness, severity and relation to study drug by cohort.
Time Frame: 0-168 days
Population: 20-60 years old, overweight and obese by BMI definition (27.5 < BMI ≤ 34.9), adult males.
Measure: Number; unit: participants
Groups:
- RZL-012 Cohort 1: A single-time injection, multiple subcutaneous injections of 40 RZL-012 administered into 8 sites (0.1mL per site):
  RZL-012: Subject receive a single-time injection. Multiple injections of RZL-012 are administered at doses of 40-180mg (8-36 injection sites, 0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 2: A single-time injection, multiple subcutaneous injections of 80mg RZL-012 administered into 16 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 40-180mg doses (8-36 injections, 0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 3: A single-time injection, multiple subcutaneous injections of 120mg RZL-012 administered into 24 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 40-180mg doses (8-36 injections, 0.1mL per site) into the abdominal subcutaneous fat.
- RZL-012 Cohort 4: A single-time injection, multiple subcutaneous injections of 180mg RZL-012 administered into 36 sites (0.1mL per site):
  Subject receive a single-time injection. Multiple injections of RZL-012 are administered at 40-180 mg (8-36 injections, 0.1mL per site) into the abdominal subcutaneous fat.
- Placebo: A single-time injection, multiple subcutaneous injections of Placebo administered into 8/16/24/36 sites (0.1mL per site)
  Placebo: Subject receive a single-time injection. Multiple injections of the Placebo are administered at 8/16/24/36 sites (0.1mL per site) into the abdominal subcutaneous fat.
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 9
participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0
  Other Adverse Events | 6 | 6 | 6 | 6 | 9
  Cardiac disorder ventricular extrasystoles | 0 | 0 | 0 | 0 | 1
  Ear and labyrinth disorders - Ear pain | 0 | 0 | 0 | 0 | 1
  Ear and labyrinth disorders Ear swelling | 0 | 0 | 0 | 0 | 1
  Ear and labyrinth disorders - Hypoacusis | 0 | 0 | 0 | 0 | 1
  Ear and labyrinth disorders otorrhoea | 0 | 0 | 0 | 0 | 2
  Aministration site condition - energy uncreased | 1 | 0 | 0 | 0 | 0
  Aministration site condition - Fatifue | 1 | 0 | 0 | 0 | 0
  Administration site condition - feeling hot | 0 | 0 | 1 | 0 | 0
  Administration site condition - bruising | 1 | 1 | 1 | 2 | 3
  Administration site condition - discolourization | 0 | 0 | 0 | 1 | 0
  Administration site condition - Erythema | 6 | 6 | 4 | 5 | 8
  Administration site condition - hemorrhage | 0 | 0 | 1 | 0 | 0
  Administration site condition - injection mass | 0 | 0 | 0 | 1 | 0
  Administration site condition - nodule | 0 | 0 | 0 | 1 | 0
  Administration site condition- Edema | 6 | 4 | 6 | 4 | 5
  Administration site condition - pain | 6 | 5 | 5 | 5 | 3
  Administration site condition- pruritus | 2 | 0 | 0 | 2 | 0
  Administration site condition - rash | 1 | 0 | 0 | 0 | 0
  Administration site condition - warmth | 2 | 0 | 0 | 0 | 0
  Administration site condition medical device reac | 0 | 0 | 1 | 0 | 0
  general condition non cardiac chest pain | 0 | 1 | 0 | 0 | 0
  Injury and procedure complications - skin abrasion | 0 | 1 | 0 | 0 | 0
  Investigations - Electrodiagram QT prolonged | 0 | 0 | 0 | 0 | 1
  Muscoloskeletal and connective tissue - myalgia | 0 | 0 | 1 | 0 | 0
  Muscoloskeletal and connective tissue - pain extre | 0 | 0 | 0 | 0 | 1
  Nervou system disorders- Dizziness | 0 | 0 | 1 | 0 | 0
  Nervou system disorders - Headache | 2 | 1 | 2 | 0 | 1
  Respeiratory, thoracic - oropharyngea pain | 0 | 0 | 1 | 0 | 0
  Respeiratory, thoracic - Respiratory tracongestion | 0 | 1 | 0 | 0 | 0
  Respeiratory, thoracic - Rhinorrhoea | 1 | 0 | 1 | 0 | 0
  skin and subcutaneous tissue disorders - erythema | 0 | 0 | 3 | 0 | 0
  skin and subcutaneous tissue disorders hyperhidros | 0 | 0 | 1 | 0 | 0
  skin and subcutaneous tissue disorders - pruritus | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Efficacy: A Significant Thermogenesis at the Injected Site.
Description: Thermogenesis is measured by thermal imaging is non-invasive, non-radiating Infra-Red thermal camera that passively measures the emitting infra-red radiation of body surface.
  Difference in temperatures between the sites (treated - not treated) by visit treatment along with the change from baseline (net-delta) in these differences by cohort and overall. Significant thermogenesis is defined as net-delta ≥ 1.
  Outcome measure data table represents the number of subjects who demonstrated an increase that is higher than 1 celsius degree.
Time Frame: 28-168 days
Measure: Count of Participants; unit: Participants
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
Participants
  Day 28 | 5 | 5 | 3 | 6 | 1
  Day 56 | 1 | 3 | 3 | 6 | 0
  Day 84 | NA — measure was not taken at this time point | NA — measure was not taken at this time point | NA — measure was not taken at this time point | 4 | 0
  Day 112 | NA — measure was not taken at this time point | NA — measure was not taken at this time point | NA — measure was not taken at this time point | 5 | 0
  Day 140 | NA — measure was not taken at this time point | NA — measure was not taken at this time point | NA — measure was not taken at this time point | 4 | 0
  Day 168 | NA — measure was not taken at this time point | NA — measure was not taken at this time point | NA — measure was not taken at this time point | 3 | 0

3. Secondary Outcome: Duration of the Thermogenic Effect From Day 28.
Description: The duration of the thermogenic effect for subjects in the active arm with thermogenic effect (net-delta ≥ 1) by visit and cohort.
Time Frame: 28-168 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
days | 5.6 (12.5) | 16.8 (15.3) | 5.6 (12.5) | 107.3 (44.9) | 0 (0)

4. Secondary Outcome: Local Reduction in Fat Mass as Measured by MRI. Local Reduction in Fat Will be Measured by Periodically MRI Scans of the Abdomen.
Description: Subcutaneous Fat Mass (SFM) ratio (treated sites / control sites) averaged over the MRI slices by visit, treatment and cohort and the change from baseline in SFM ratio (in % from the ratio at baseline) compared between the treatment arms.
Time Frame: 28-168 days
Population: In cohort 4, one subjects was not analyzed due to MRI image quality (bubble)
Measure: Mean (Standard Deviation); unit: percentage of SFM reduction
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 7
percentage of SFM reduction
  Day 28 | -0.62 (5.17) | -9.15 (10.55) | -9.1 (4.27) | -14.68 (8.16) | 2.94 (10.08)
  Day 56 | NA (NA) — Measurement was not perform at this time point for cohort 1 subjects | -8.56 (8.85) | -10.52 (8.42) | -18.10 (10.93) | 3.61 (3.48)
  Day 84 | NA (NA) — Measurement was not perform at this time point for cohort 1 subjects | NA (NA) — Measurement was not perform at this time point for cohort 2 subjects | NA (NA) — Measurement was not perform at this time point for cohort 3 subjects | -12.75 (9.83) | -6.57 (9.78)
  Day 112 | NA (NA) — Measurement was not perform at this time point for cohort 1 subjects | NA (NA) — Measurement was not perform at this time point for cohort 2 subjects | NA (NA) — Measurement was not perform at this time point for cohort 3 subjects | -16.10 (13.81) | -8.2 (11.54)
  Day 140 | NA (NA) — Measurement was not perform at this time point for cohort 1 subjects | NA (NA) — Measurement was not perform at this time point for cohort 2 subjects | NA (NA) — Measurement was not perform at this time point for cohort 3 subjects | -12.46 (11.26) | -2.9 (0.45)
  Day 168 | NA (NA) — Measurement was not perform at this time point for cohort 1 subjects | NA (NA) — Measurement was not perform at this time point for cohort 2 subjects | NA (NA) — Measurement was not perform at this time point for cohort 3 subjects | -14.32 (10.94) | -2.54 (8.57)
Statistical Analysis 1: Comparison: RZL-012 Cohort 1 vs Placebo; The Kruskal-Wallis T-test was applied for analyzing the difference in between the study groups; Test type: Superiority; p > 0.05, Kruskal-Wallis
Statistical Analysis 2: Comparison: RZL-012 Cohort 2 vs Placebo; The Kruskal-Wallis T-test was applied for analyzing the difference in between the study groups, at day 28 and Day 56; Test type: Superiority; p < 0.05, Kruskal-Wallis
Statistical Analysis 3: Comparison: RZL-012 Cohort 3 vs Placebo; The Kruskal-Wallis T-test was applied for analyzing the difference in between the study groups; Test type: Superiority; p < 0.05, Kruskal-Wallis
Statistical Analysis 4: Comparison: RZL-012 Cohort 4 vs Placebo; The Kruskal-Wallis T-test was applied for analyzing the difference in between the study groups; Test type: Superiority; p < 0.05, Kruskal-Wallis

5. Secondary Outcome: Changes in Fasting Blood Glucose From Baseline.
Description: Changes from baseline in fasting blood glucose by visit, treatment, and cohort.
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
mg/dL
  Day -1 | 86.7 (4.2) | 91.3 (5.16) | 91.7 (7.47) | 90.8 (7.17) | 93.2 (3.93)
  Day 56 | 93 (3.22) | 92.8 (11.8) | 93.3 (7.58) | 93.7 (5.3) | 94.6 (6.6)
Statistical Analysis 1: Comparison: RZL-012 Cohort 1 vs Placebo; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: RZL-012 Cohort 2 vs Placebo; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: RZL-012 Cohort 3 vs Placebo; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: RZL-012 Cohort 4 vs Placebo; Test type: Other; p > 0.05, t-test, 2 sided

6. Secondary Outcome: Changes in Blood Lipid Profile From Baseline.
Description: Changes from baseline in lipid profile by visit, treatment, and cohort.
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
mg/dL
  Cholesterol Day -1 | 188 (32.8) | 199 (11) | 196 (41.4) | 170.8 (23) | 186.7 (19.8)
  Cholesterol Day 56 | 184 (39.8) | 205 (29.7) | 201.7 (46.1) | 176 (28.6) | 182.4 (19.3)
  HDL Day -1 | 43.5 (7.23) | 44.33 (11.1) | 41.5 (6) | 44 (6.87) | 42.44 (5.6)
  HDL Day 56 | 40 (9.44) | 50.8 (14.2) | 41.5 (9.9) | 45.3 (5.05) | 41.14 (7)
  LDL Day -1 | 129 (33.5) | 126.5 (13.3) | 134 (33) | 105.5 (15) | 116 (10.3)
  LDL Day 56 | 120 (31.3) | 132 (23.9) | 134.7 (37) | 128 (0) | 103 (14.8)
  Triglycerides Day -1 | 107.3 (42.3) | 131 (77) | 112.5 (58.9) | 121.7 (39.3) | 155.8 (98)
  Triglycerides Day 56 | 118 (85.4) | 136 (61.1) | 193.5 (16.7) | 128.33 (55.4) | 234 (220)

7. Secondary Outcome: Pharmacokinetics: Establishing Pharmacokinetic Profile of RZL-012.
Description: Averaged Cmax values by cohort.
Time Frame: 1-2 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 84.15 (16.27) | 181.89 (49.86) | 241 (72.09) | 344 (73.7)

8. Secondary Outcome: Changes in Body Weight
Description: Changes from baseline in body weight by visit, treatment, and cohort.
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
Kg
  Weight Day -1 | 103.3 (11.1) | 95.4 (6.9) | 101.3 (20.3) | 96.1 (12.6) | 99.1 (8.1)
  Weight Day 56 | 104.4 (12.5) | 96.1 (7.8) | 103.4 (22.4) | 96 (12.3) | 101.2 (9.7)

9. Secondary Outcome: Changes in Waist to Hip Ratio [WHR]
Description: Changes from baseline in WHR by visit, treatment, and cohort. WHR is calculated by measurements of waist circumference and hip circumference.
Time Frame: 56 days
Measure: Mean (Standard Error); unit: ratio
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
ratio
  Waist to hip ratio Day -1 | 1 (0.1) | 1 (0) | 1 (0.1) | 1 (0) | 1 (0.1)
  Waist to hip ratio Day 56 | 1 (0) | 1 (0) | 1 (0) | 1 (0) | 1 (0.1)

10. Secondary Outcome: Elucidation of the Histological Changes Account for the Thermogenic Effect.
Description: An abdominal subcutaneous adipose tissue biopsy will be taken from the injected side.
  Histology results will be assessed for 2 subjects who were injected with 120 mg RZL-012 and for one subject who was injected with placebo.
Time Frame: 56 days
Population: Biopsy was done only for 2 active and 1 placebo subjects in cohort 3. Biopsy was not done in subjects from cohorts 1,2 or 4.
Measure: Count of Participants; unit: Participants
Arm/Group | RZL-012 Cohort 3 | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

11. Secondary Outcome: Change From Baseline in Inflammatory Markers and Cytokines. Testing of Inflammatory Markers and Cytokines Will be Conducted by Blood Sampling.
Description: Changes from baseline in inflammatory markers and cytokines by visit, treatment, and cohort.
  Testing of inflammatory markers and cytokines will be conducted by blood sampling.
Time Frame: 28 days
Population: The study was designed in a way that inflammation marker will be measured only for active and placebo subjects from cohorts 2-4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5
mg/dL
  CRP Day -1 (mg/dL) | 0.2 (0.13) | 0.6 (1.08) | 0.5 (0) | 0.2 (0.1)
  CRP Day 28 (mg/dL) | 0.27 (0.31) | 0.2 (0.12) | 0.43 (0.15) | 0.2 (0.1)
Statistical Analysis 1: Comparison: RZL-012 Cohort 4 vs Placebo; Test type: Other; p > 0.05, t-test, 2 sided

12. Secondary Outcome: Pharmacokinetics: Establishing Pharmacokinetic Profile of RZL-012.
Description: Averaged Tmax values by cohort.
Time Frame: 0.5, 1,2,3,4,5,6,8,12,16,24,30 hours
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hour | 1.83 (0.41) | 1.83 (0.41) | 1.83 (0.41) | 2 (0)

ADVERSE EVENTS:
Time Frame: All reported adverse events were coded to a standard set of terms using MedDRA coding dictionary. Cohort 4 subjects were followed up for Adverse Events up to 168 days following injection.
Description: None of the subjects was reported with SAEs. None of the subjects died during the study
Arm/Group | RZL-012 Cohort 1 | RZL-012 Cohort 2 | RZL-012 Cohort 3 | RZL-012 Cohort 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RZL-012 Cohort 1 (N=6) | RZL-012 Cohort 2 (N=6) | RZL-012 Cohort 3 (N=6) | RZL-012 Cohort 4 (N=6) | Placebo (N=9)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ear swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Energy increased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site Erythema (General disorders) | 6 (6) | 6 (7) | 4 (5) | 5 (7) | 8 (11)
Injection site hemmorhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site Edema (General disorders) | 6 (7) | 4 (4) | 6 (7) | 4 (5) | 5 (6)
Injection site pain (General disorders) | 6 (6) | 5 (5) | 5 (8) | 5 (6) | 3 (3)
Injection site pruritus (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiac QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Orpharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT03171415/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03171415/SAP_001.pdf